CLINICAL TRIAL: NCT07313670
Title: Outcome of Using Hydrocortisone in Early Treatment of Pediatric Septic Shock
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-JAWARIA-KARACHI
Record Dates: First submitted 2025-12-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone Group (Experimental): Children will receive early intravenous hydrocortisone at 2 mg/kg/day divided every 6 hours, continued for 7 days or until resolution of shock.
  Interventions: Drug: Intravenous Hydrocortisone; Drug: Standard care
- Standard Care Group (Experimental): The children will be managed by following standard institutional treatment protocol.
  Interventions: Drug: Standard care

INTERVENTIONS:
Drug: Intravenous Hydrocortisone — Children will receive early intravenous hydrocortisone at 2 mg/kg/day divided every 6 hours, continued for 7 days or until resolution of shock.
  Arms: Hydrocortisone Group
Drug: Standard care — The children will be managed by following standard institutional treatment protocol.

SUMMARY:
Although, hydrocortisone has shown promise in managing refractory shock, its role in early septic shock management remains unclear. This study aims to provide robust evidence on the clinical and hemodynamic outcomes of early hydrocortisone use in pediatric septic shock, contributing to standardized treatment protocols and improved survival rates.

DETAILED DESCRIPTION:
Despite global advancements in pediatric critical care, mortality and morbidity in septic shock remain unacceptably high. Although data suggest a reduction in mortality with steroid therapy in refractory shock, specific data for hydrocortisone in pediatrics are limited. The findings of this study would not only be a valuable addition to the existing stats but might also help develop a protocol for the use of hydrocortisone therapy in children with septic shock, seeking an earlier recovery from organ failure, earlier reversal of shock, and lower mortality in children with sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Children of any gender
* Aged 2 month to 12 years
* Diagnosed with septic shock
* Admitted to the pediatric intensive care unit

Exclusion Criteria:

* Known adrenal insufficiency or congenital adrenal hyperplasia
* History of corticosteroid use within the past 7 days
* Terminal illness or "do-not-resuscitate (DNR)" status
* Severe immunocompromise (e.g., advanced malignancy, HIV stage IV)
* Known allergy to hydrocortisone

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  The mortality will be labeled 'yes' if a patient dies within 28 days of admission.

SECONDARY OUTCOMES:
Duration of vasopressor | 28 days
  Vasopressor therapy time will be computed from the start of treatment until hemodynamic stability is attained.
Length of pediatric intensive care unit stay | 28 days
  The time will be calculated from admission in the pediatric intensive care unit until discharge or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Jawaria Ibrahim, Principal Investigator — Abbasi Shaheed Hospital; Ibrahim Shakoor, FCPS, Study Director — Abbasi Shaheed Hospital
Locations (1):
- Abbasi Shaheed Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.